CLINICAL TRIAL: NCT03103399
Title: A Multicentre, Double-blind, Randomised, Active- and Placebo-controlled Trial to Investigate the Efficacy and Tolerability of Nebicapone in Parkinson's Disease Patients With "Wearingoff" Phenomenon Treated With Levodopa/Carbidopa or Levodopa/Benserazide
Brief Title: Efficacy and Tolerability of Nebicapone in Parkinson's Disease Patients With "Wearingoff" Phenomenon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-202
Record Dates: First submitted 2017-03-28; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone; nebicapone; Levodopa; Benserazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 50 mg nebicapone (Experimental): At Visit V2, patients received a supply of a placebo to take concomitantly with each levodopa/DDCI dose for the duration of the run-in period (Period 1). At the end of Period 1, patients were randomised to receive 50 mg of the study treatment in addition to their levodopa/DDCI therapy for the duration of the double-blind (Period 2)
  Interventions: Drug: Nebicapone; Drug: Levodopa/DDCI; Drug: Placebo
- 100 mg nebicapone (Experimental): At Visit V2, patients received a supply of a placebo to take concomitantly with each levodopa/DDCI dose for the duration of the run-in period (Period 1). At the end of Period 1, patients were randomised to receive 100 mg of the study treatment in addition to their levodopa/DDCI therapy for the duration of the double-blind (Period 2)
  Interventions: Drug: Nebicapone; Drug: Levodopa/DDCI; Drug: Placebo
- 150 mg nebicapone (Experimental): At Visit V2, patients received a supply of a placebo to take concomitantly with each levodopa/DDCI dose for the duration of the run-in period (Period 1). At the end of Period 1, patients were randomised to receive 150 mg of the study treatment in addition to their levodopa/DDCI therapy for the duration of the double-blind (Period 2)
  Interventions: Drug: Nebicapone; Drug: Levodopa/DDCI; Drug: Placebo
- 200 mg entacapone (Active Comparator): At Visit V2, patients received a supply of a placebo to take concomitantly with each levodopa/DDCI dose for the duration of the run-in period (Period 1). At the end of Period 1, patients were randomised to receive 200 mg of entacapone (Comtan®) in addition to their levodopa/DDCI therapy for the duration of the double-blind (Period 2)
  Interventions: Drug: Comtan®; Drug: Levodopa/DDCI; Drug: Placebo
- Placebo (Placebo Comparator): At Visit V2, patients received a supply of a placebo to take concomitantly with each levodopa/DDCI dose for the duration of the run-in period (Period 1). At the end of Period 1, patients were randomised to receive study treatment matching placebo tablets in addition to their levodopa/DDCI therapy for the duration of the double-blind (Period 2)
  Interventions: Drug: Levodopa/DDCI; Drug: Placebo

INTERVENTIONS:
Drug: Comtan® — 200 mg entacapone were to be taken concomitantly with each levodopa/DDCI dose.
  Other Names: entacapone
  Arms: 200 mg entacapone
Drug: Nebicapone — 50 mg, 100 mg and 150 mg doses of nebicapone were to be taken concomitantly with each levodopa/DDCI dose.
  Other Names: BIA 3-202
  Arms: 100 mg nebicapone; 150 mg nebicapone; 50 mg nebicapone
Drug: Levodopa/DDCI — Prior to the study, all patients were to have been receiving levodopa/DDCI therapy for at least 1 year with clear clinical improvement. At entry to the study, patients were to be receiving levodopa/DDCI therapy of at least 4 but not more than 8 (inclusive) standard daily doses.
  All patients were to continue receiving levodopa/DDCI during the study. Levodopa and DDCI were prescribed by the investigators and purchased locally by patients.
  Other Names: Levodopa plus a dopa decarboxylase inhibitor (DDCI: carbidopa or benserazide)
Drug: Placebo — Administered orally as encapsulated tablets, which were identical in appearance to the study drugs
  Other Names: placebo tablets

SUMMARY:
The purpose of this study was to investigate the effect on the "wearing-off" phenomenon of 3 different doses of nebicapone (NEB 50 mg, 100 mg and 150 mg), compared with entacapone and placebo when dministered concomitantly with existing treatment with levodopa plus a dopa decarboxylase inhibitor (DDCI: carbidopa or benserazide).

DETAILED DESCRIPTION:
The study was conducted in 40 sites in Europe and South America: Argentina (6); Austria (2); Brazil (5); France (1); Hungary (4); Poland (7); Portugal (2); Romania (7); and Ukraine (6).

Multicentre study with a screening visit (Visit V1), a single-blind placebo run-in period of 1 or 2 weeks (Period 1, Visits V2 to V3), and an 8-week randomised, double-blind, activeand placebo-controlled, parallel-group (5 groups) treatment period (Period 2, Visits V3 to V7). In Hungary only: a 1-week tapering-off period was added by amendment #1HU. The dosage of nebicapone was to be tapered off stepwise during 6 days. This period was to end with a follow-up Visit V8.

ELIGIBILITY:
Inclusion Criteria:

At Visit V1 (screening), patients had to be/have:

* Ability to comprehend and willingness to sign an informed consent form
* Aged 30 to 80 years, inclusive
* Diagnosis of idiopathic Parkinson's disease according to the Brain Bank Clinical Diagnosis Criteria of the UK Parkinson's Disease Society [Hughes et al, 1992]
* Disease severity less than Stage 5 (modified Hoehn & Yahr staging) while during the "off" time
* Treated with levodopa plus DDCI for at least 1 year with clear clinical improvement
* Treated with 4 to 8 (inclusive) daily doses of standard levodopa plus DDCI (bedtime dose of a slow-release formulation is permitted)
* Stable regimen of levodopa plus DDCI and other anti Parkinson drugs for at least 4 weeks before screening
* Signs of end-of-dose "wearing-off" phenomenon (end-of-dose deterioration) with average total daily "off" time while awake of at least 1.5 hours excluding the early morning pre first dose "off" period despite optimal anti Parkinson therapy, determined subjectively and objectively (observations of the investigator) for a minimum of 2 months before screening
* Ability to keep reliable diaries of motor fluctuations (alone or with family/caregiver assistance)
* Patient must be amenorrhoeic for at least 1 year or surgically sterile for at least 6 months before screening. In case of women of childbearing potential, patient must be using double-barrier contraceptive method.

At Visit V2 (entry to Period 1), patients had to have the results of laboratory tests acceptable by the investigator (not clinically relevant for the well being of the patient or for the purpose of the study).

At Visit V3 (randomisation), patients had to have:

* At least 80% treatment medication (levodopa/DDCI plus investigational product) compliance with the recommended dosage regimen during Period 1
* Self-rating diary charts filled in in accordance with the diary chart instructions; less than 3 errors per day are allowed
* Average of at least 1.5 "off" hours per day (excluding the early morning pre first dose "off" period) on the 3 day diaries, filled in on the 3 days preceding Visit V3, according to the self-rating diary charts completed during Period 1

Exclusion Criteria:

At Visit V1 (screening), patients were not to be/have:

* Non-idiopathic Parkinson's disease (atypical parkinsonism, symptomatic parkinsonism, Parkinson-plus syndrome)
* Dyskinesia disability score more than 3 in the Unified Parkinson's Disease Rating Scale (UPDRS) IV.A item 33
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criterion for dementia
* Major depressive episode within the 6 months before screening
* Treatment with entacapone, tolcapone, neuroleptics, antidepressants (except serotonin-specific reuptake inhibitors or imipraminics [desipramine, imipramine, clomipramine and amitriptyline]), monoamine oxidase inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation or rasagiline up to 1 mg/day), or antiemetics (except domperidone) within the 3 months before screening
* Treatment with apomorphine within the previous month before screening
* Dosage change of concomitant anti Parkinson medication within 4 weeks of screening
* Any investigational product within the 3 months (or within 5 half-lives, whichever is longer) before screening
* A psychiatric or any medical condition that might place the patient at increased risk or interfere with assessment
* A clinically relevant electrocardiogram (ECG) abnormality
* A history or current evidence of heart disease, including but not limited to myocardial infarction, angina, congestive heart failure and cardiac arrhythmia
* Phaeochromocytoma
* Known hypersensitivity to the ingredients of products used
* Unstable concomitant disease being treated with changing doses of medication
* History or current evidence of any relevant disease in the context of this study, i.e. with respect to the safety of the patient or related to the study conditions, e.g. that may influence the absorption or metabolism (e.g. hepatic impairment) of the investigational drug
* Any abnormality in the liver enzymes above 2 times the upper limit of the normal range

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-09-26 (Actual); Primary Completion 2007-09-21 (Actual); Study Completion 2007-09-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in absolute "off" time (time with poor mobility or complete immobility) at Visit V7 | 8 weeks
  Baseline values for all efficacy variables were the values from Visit V3, and change from baseline refers to absolute change from baseline at Visit 7 (end of the 8-week treatment period)

SECONDARY OUTCOMES:
Proportion of "off" time responders | 8 weeks
  "off" time responders are defined as patients with a reduction of at least 1 hour in absolute "off" time since baseline (Visit V3).
Proportion of "on" time responders | 8 weeks
  "on" time responders are defined as patients with an increase of at least 1 hour in absolute total "on" time since baseline (Visit V3).

IPD SHARING:
Plan to Share IPD: Undecided